CLINICAL TRIAL: NCT02441010
Title: Application of Monitoring and Intervention Technologies in Suboptimal Health Status in a General Population in China
Brief Title: Application of Monitoring and Intervention Technologies in Suboptimal Health Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qiang Zeng, MD, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012BAI37B04-05
Record Dates: First submitted 2015-05-01; First posted 2015-05-12 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Suboptimal Health Status; Metabolic Abnormality
MeSH Terms: interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group 1 (No Intervention): Participants without suboptimal health status are randomly grouped into the group without monitor (Group 1) and the monitor group (Group 2 or Group 3). Thus, no monitoring or intervention technologies are used in Group 1.
- Group 2 (Sham Comparator): Group 2 are participants without metabolic abnormality in the monitor group. Group 2 use the monitoring device with three months.
  Interventions: Device: monitoring device
- Group 3 (Sham Comparator): Group 3 are participants with metabolic abnormality in the monitor group. Group 3 use the monitoring device and the health information push technology with three months.
  Interventions: Other: health information push technology; Device: monitoring device
- Group 4 (Active Comparator): All of participants with suboptimal health status use the monitoring device with three months, and are randomly grouped into the non-intervention group (Group 4 or Group 5) and the intervention group using the meridian therapy instrument (Group 6 or Group 7). Group 4 are participants without metabolic abnormality in the non-intervention group. No intervention technologies are used in Group 4.
  Interventions: Device: monitoring device
- Group 5 (Active Comparator): Group 5 are participants with metabolic abnormality in the non-intervention group. Group 5 use the health information push technology with three months.
  Interventions: Other: health information push technology; Device: monitoring device
- Group 6 (Experimental): Group 6 are participants without metabolic abnormality in the intervention group. Group 6 use the meridian therapy instrument with two weeks. If the suboptimal health status is not improved, then the meridian therapy instrument will continue to be used with an interval of one week.
  Interventions: Device: meridian therapy instrument; Device: monitoring device
- Group 7 (Experimental): Group 7 are participants with metabolic abnormality in the intervention group. Group 7 use the health information push technology with three months and the meridian therapy instrument with two weeks. Similar with Group 6, if the suboptimal health status is not improved after the treatment of the meridian therapy instrument, then the instrument will continue to be used with an interval of one week.
  Interventions: Device: meridian therapy instrument; Other: health information push technology; Device: monitoring device

INTERVENTIONS:
Device: meridian therapy instrument — The meridian therapy instrument are widely used to improve the physical and relieve fatigue and pain in many hospitals by the field-effect.
  Other Names: KangRu
  Arms: Group 6; Group 7
Other: health information push technology — The health information push technology regularly send health information on the measurements of body weight control and the improvement of a healthy lifestyle.
  Other Names: Health Management System
  Arms: Group 3; Group 5; Group 7
Device: monitoring device — The monitoring device is used to monitor a person's blood pressure, blood glucose, oxygen saturation, body weight, and energy consumption by Bluetooth Wireless technology.
  Other Names: BianQueFeiJiu
  Arms: Group 2; Group 3; Group 4; Group 5; Group 6; Group 7

SUMMARY:
The purpose of this study is to use monitoring and intervention technologies in suboptimal health status in a general population in China and evaluate the effectiveness of these technologies in the improvement of suboptimal health status.

DETAILED DESCRIPTION:
The Suboptimal health status questionnaire (SHSQ-25) is used to evaluate the suboptimal health status. The SHSQ-25 includes 25 questions. The score of the SHSQ-25 is from 0 to 100. Suboptimal health status is defined as the SHSQ-25 score above than 35. The higher scores of the SHSQ-25 one gets, the more severity of suboptimal health status he/she has. All participants are asked to fill in the SHSQ-25 before and after the intervention. If the score decreases after the intervention, it means that the suboptimal health status has been improved.

A monitoring device is used to monitor a person's blood pressure, blood glucose, oxygen saturation, body weight, and energy consumption by Bluetooth Wireless technology. Intervention technologies include a health information push technology and a field-effect meridian therapy instrument.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 60 years.
2. written informed consent.

Exclusion Criteria:

1. history of system diseases, such as cardiovascular diseases, digestive system diseases, diseases of respiratory system, blood and immune system diseases, nervous system diseases, endocrine system diseases, and diseases of the genitourinary system.
2. history of mental illness.
3. pregnant or breastfeeding.
4. use of antihypertensive, antidiabetic, or lipid-lowering drugs within the past two weeks.
5. participation in another trial.
6. unable to promise to not use drugs and other fish oils during the study.
7. unable to provide informed written consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2014 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
the improvement of suboptimal health status | three months
  The improvement of suboptimal health status is evaluated by the change of the SHSQ-25 scores after intervention.

SECONDARY OUTCOMES:
the change of metabolic abnormality | three months
  To investigate the change of metabolic abnormality when the monitoring and/or intervention technologies are used. The definition of metabolic abnormality is met when one or more of the following criteria are present: (1) blood pressure ≥ 130 mmHg; (2) fasting blood glucose ≥ 100 mg/dl; (3) body mass index ≥ 28 kg/m2; (4) dyslipidemia (total cholesterol ≥ 200 mg/dl, triglyceride ≥ 150 mg/dl, low-density lipoprotein cholesterol ≥ 130 mg/dl, and/or high-density lipoprotein cholesterol < 40 mg/dl).

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zeng, M.D, Study Chair — Chinese PLA General Hospital; Song Leng, M.D, Principal Investigator — The Second Affiliated Hospital of Dalian Medical University; Sheng-Yong Dong, M.D., Ph.D, Principal Investigator — General Staff Department of PLA
Locations (2):
- China (2):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning